CLINICAL TRIAL: NCT06426277
Title: Effectiveness of the Diabetes Prevention Program on the Incidence of Type 2 Diabetes Mellitus Among Brazilian Individuals: Randomized Clinical Trial (PROVEN-DIA Study)
Brief Title: Effectiveness of the Brazilian Diabetes Prevention Program
Acronym: PROVEN-DIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROVEN-DIA ECR
Record Dates: First submitted 2024-03-19; First posted 2024-05-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Prediabetic State; Pre Diabetes
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brazilian Diabetes Prevention Program (face-to-face care) (Experimental): The PROVEN-DIA program is a structured lifestyle change initiative organized into modules that include nutrition, physical activity, and self-care. Based on materials already made available by the Brazilian Ministry of Health, such as the Dietary Guidelines for the Brazilian Population and the Physical Activity Guide for the Brazilian Population, we developed a protocol that considers health status, lifestyle habits, and motivation to set lifestyle change goals.
  Specifically, in this arm of the study, PROVEN-DIA will be delivered through in-person individual and group sessions, as well as virtual interactions with coaches/facilitators.
  There will be 23 in-person visits and 15 virtual contacts.
  Interventions: Behavioral: Brazilian Diabetes Prevention Program (face-to-face care)
- Brazilian Diabetes Prevention Program (remote care) (Active Comparator): The PROVEN-DIA program is a structured lifestyle change initiative organized into modules that include nutrition, physical activity, and self-care. Based on materials already made available by the Brazilian Ministry of Health, such as the Dietary Guidelines for the Brazilian Population and the Physical Activity Guide for the Brazilian Population, we developed a protocol that considers health status, lifestyle habits, and motivation to set lifestyle change goals.
  Specifically, in this arm of the study, PROVEN-DIA will be delivered 100% virtual.
  There will be 38 virtual contacts.
  Interventions: Behavioral: Brazilian Diabetes Prevention Program (remote care)
- Control Group (Active Comparator): Nutritional guidance is based on the Dietary Guidelines for the Brazilian Population, and physical activity recommendations follow the Physical Activity Guide for the Brazilian Population. In other words, this group uses the same tools to guide patients as the PROVEN-DIA intervention. However, it is not structured as a program with a protocol to help professionals set lifestyle change goals with patients. This group simulates the current standard of care in primary healthcare in Brazil.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Brazilian Diabetes Prevention Program (face-to-face care) — A Program structured in 28 visits (in group and individual) and 21 contacts (through phone calls or video calls) to guide the improvement of diet quality, self-care, and regular practice of physical activity
  Arms: Brazilian Diabetes Prevention Program (face-to-face care)
Behavioral: Diet — Hypocaloric diet prescription
  Arms: Control Group
Behavioral: Brazilian Diabetes Prevention Program (remote care) — A Program structured in 49 contacts delivered through telehealth (through phone calls or video calls between professional and participant) to guide the improvement of diet quality, self-care, and regular practice of physical activity
  Arms: Brazilian Diabetes Prevention Program (remote care)

SUMMARY:
The aim of this multicenter, randomized controlled trial is to assess the effectiveness of the Brazilian Diabetes Prevention Program (delivered face-to-face or via e-health) in preventing type 2 diabetes (T2D) in at least 1,590 adults at high risk of T2D over a 3-year follow-up period. Our outcomes include the incidence of T2D, body weight (kg), BMI, glycemic biomarkers, use of antidiabetic drugs, the proportion of individuals achieving controlled glycemia or HbA1c levels without medication, diet quality, moderate-to-vigorous physical activity (min/week), prevalence of physical inactivity, sleep quality, perceived stress, alcohol consumption, smoking, and quality of life. In addition, social, cultural, educational, and geographical factors at the community level will be analyzed throughout the follow-up to determine their association with the incidence of T2D.

DETAILED DESCRIPTION:
This is a multicenter controlled randomized trial coordinated by the Hospital Beneficência Portuguesa in São Paulo-Brazil and made possible by PROADI-SUS (SUS Institutional Development Support Program).

ELIGIBILITY:
Inclusion Criteria

* Be 18 years or older (no maximum age for being eligible)
* Have a body mass index (BMI) between 25 and 34,9kg/m²
* Have, at least, one electronic device (includes any of the following devices):

  * Computer
  * Laptop/notebook
  * Tablet
  * Smartphone
* Have access to internet (broadband, 3G, 4G, 5G, among others) Without previous nutritional counseling (within the 6 months prior to recruitment/randomization/intervention) Without supervision by a Physical Education Professional (Personal Trainer) in the past 6 months
* Living near the research center (at maximum 60 minutes)
* Had a blood test result in the prediabetes range within the last three months prior to the recruitment/randomization/intervention (includes any of these tests and results):

  * Hemoglobin levels (HbA1c): 5.7-6.4%
  * Blood glucose 2 hours after an oral glucose tolerance: 140-199 mg/dL

Exclusion Criteria:

* Diagnosis of Diabetes Mellitus
* Underlying disease likely to limit life expectancy and/or increase the risk of interventions influencing the risk of developing T2D
* Diagnosis of Renal Disease
* Diagnosis of Pulmonary Disease
* Gastrointestinal Disease
* Secondary prevention for Cardiovascular Disease
* Endocrine Diseases
* Weight loss exceeding 10% in the last 6 months (except postpartum-related)
* Uncontrolled Hypertension
* Diagnosis of Polycystic Ovary Syndrome (self-reported)
* Patients undergoing treatment for Tuberculosis
* Presence of diseases that may severely reduce life expectancy or the ability to participate in the study
* Pregnant or breastfeeding women
* Severe psychiatric disorders that, in the opinion of the clinical team, hinder participation in the program
* Acute or chronic excessive alcohol consumption
* Congestive Heart Failure (CHF) with a New York Heart Association Functional Class (NYHA) > 2
* Need for referral to a cardiologist according to the Physical Activity Readiness Questionnaire (PAR-Q)
* Current or recent participation (within the last six months) in another clinical trial that impacts the interventions and/or is associated with the study outcomes (in case of doubt, contact the coordinating center)
* Likely relocation away from the research collaborating center within the next 3 years
* Another household member is a participant or a team member of the PROVEN-DIA study
* Unwillingness to accept treatment assignment by randomization and/or refusal to participate in the study (signing the Informed Consent Form)
* Continuous use of the following medications:

Corticosteroids other than topical, ophthalmic, or inhaled preparations Antineoplastic agents Psychoactive agents Other medications.

• Participant from the pilot Randomized Clinical Trial (Brazilian Diabetes Prevention Program: Pilot Study (PROVEN-Dia), NCT05689658)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes mellitus (T2DM) | 36 months
  to analyze the incidence of type 2 diabetes mellitus

SECONDARY OUTCOMES:
Mean value of Glycated Hemoglobin level (HbA1c in %) | 6, 12, 24 and 36 months
  to compare mean HbA1c(%) obtained through laboratory exams/tests between groups
Mean value of Fasting Blood Glucose (mg/dL) | 6, 12, 24 and 36 months
  to compare mean fasting blood glucose (mg/dL) obtained through laboratory exams/tests between groups
Number of Participants with controlled Fasting blood glucose (<126mg/dL) | 6, 12, 24 and 36 months
  to compare the proportion of individuals with controlled blood glucose (<126mg/dl) obtained through laboratory exams/tests without the use of hypoglycemic medication
Number of Participants with controlled Glycated Hemoglobin level (<6.4%) | 6, 12, 24 and 36 months
  to compare the proportion of individuals with HbA1c (<6.4%) obtained through laboratory exams/tests without the use of hypoglycemic medication
body weight | 6, 12, 24 and 36 months
  to compare mean weight (kg) between groups
Number of Participants who performed, at least, 150 minutes of moderate-to-vigorous physical activity obtained by International Physical Activity Questionnaire short form | 6, 12, 24 and 36 months
  to compare the proportion of individuals who are physically active (>150 minutes of moderate to vigorous physical activity) and inactive (<150 minutes of moderate to vigorous physical activity) between groups
Minutes spent on moderate-to-vigorous physical activity | 6, 12, 24 and 36 months
  to compare mean time in minutes of practice of moderate/vigorous physical activity over a week between groups
Moderate-to-vigorous physical activity and sedentary behavior | 6, 12, 24 and 36 months
  to compare the proportion of individuals engaging in moderate or vigorous physical activity and sedentary behavior
Physical activity | 6, 12, 24 and 36 months
  to compare the proportion of individuals who engage in 150 minutes or more of physical activity per week
Sedentary behavior | 6, 12, 24 and 36 months
  to compare the proportion of sedentary individuals
Quality of diet (Mean score of The Diet Quality Index Revised (DQI-R)) | 6, 12, 24 and 36 months
  to compare mean score of the Diet Quality Index Revised (DQI-R) between groups Minimum: 0 Maximum: 100 When higher the score, better the quality of diet
Mean of kcal from ultra processed food intake | 6, 12, 24 and 36 months
  to compare the mean caloric intake (kcal) from ultra-processed foods obtained through two 24-hour Dietary Recall applied within a period of fifteen days
Delta value (Change score from baseline to 6, 12, 24 and 36 months) for each domain of Quality of life obtained through Short Form Health Survey (SF-36) | 6, 12, 24 and 36 months
  to analyze the quality of life based on delta value of the eight domains (Functional capacity, Physical aspects, Pain, General health status, Vitality, Social aspects, Emotional aspects and Mental health) When higher the score, better the quality of life related to the assessed domain
Cost | 36 months
  To compare the cost of interventions. To estimate healthcare system costs, we will consider only direct medical costs, which include screening costs, intervention costs, and costs of healthcare service utilization. To estimate social costs, we will consider not only direct medical costs but also non-medical direct costs, such as transportation, food, and accommodation expenses reported by participants when seeking medical assistance, as well as time spent traveling to and participating in group sessions. Additionally, we will include indirect costs, calculated based on the assumption that each necessary hospitalization results in a loss of 9 hours of paid work and each outpatient visit results in a loss of half a day (4.5 hours) of paid work
Scholarity | 36 months
  To analyze the correlation between years of study and the incidence of type 2 diabetes
Geo-Stratified Analysis | 36 months
  T2DM incidence across Brazillian five geographic regions (South, Southeast, Midwest, West, and Northwest)
Household income | 36 months
  Association between T2DM incidence and individual Low or high income (accessed by ABEP - Critério Brasil 2022 questionnaire. A Brazilian validated questionnaire to evaluate Household income)
Neighbourhood value | 36 months
  correlation between neighborhood value (as assessed using the Gini index) and incidence of type 2 diabetes (DM2)
Mean value of BMI (kg/m2) | 6, 12, 24 and 36 months
  to compare mean BMI (kg/m2) between groups
Number of Participants in use of hypoglycemic medication | 6, 12, 24 and 36 months
  to compare the proportion of individuals in use of hypoglycemic medication
delta body weight | 6, 12, 24 and 36 months
  to compare mean delta weight (kg) between groups (delta = final mean weight - baseline mean weight)
delta glycemia | 6, 12, 24 and 36 months
  To compare the mean delta glycemia (mg/dL) between groups:
  Delta = Mean glycemia at the final measurement - Mean glycemia at baseline
  This approach evaluates the difference in blood glucose changes across the groups over the study period, reflecting the intervention's impact on glycemic control.
delta HbA1c (%) | 6, 12, 24 and 36 months
  To compare the mean delta HbA1c (%) between groups:
  Delta = Mean HbA1c at the final measurement - Mean HbA1c at baseline
  This approach evaluates the difference in blood glucose changes across the groups over the study period, reflecting the intervention's impact on glycemic control.
delta Insulin (μU/mL) | 6, 12, 24 and 36 months
  To compare the mean delta Insulin (μU/mL) between groups:
  Delta = Mean Insulin at the final measurement - Mean Insulin at baseline
  This approach evaluates the difference in Insulin changes across the groups over the study period, reflecting the intervention's impact on glycemic control.
delta HOMA-IR (homeostasis model assessment-estimated insulin resistance) | 6, 12, 24 and 36 months
  To compare the mean delta HOMA-IR between groups:
  Delta = Mean HOMA-IR at the final measurement - Mean HOMA-IR at baseline
  HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is calculated using the following formula:
  HOMA-IR = [Fasting insulin (μU/mL) × Fasting glucose (mg/dL)] / 405
  This approach evaluates the difference in insulin resistance changes across the groups over the study period, reflecting the intervention's impact on metabolic control.
delta HOMA-Beta *homeostasis model assessment of β-cell function) | 6, 12, 24 and 36 months
  To compare the mean delta HOMA-Beta between groups:
  Delta = Mean HOMA-Beta at the final measurement - Mean HOMA-Beta at baseline
  HOMA-Beta (Homeostatic Model Assessment of Beta-Cell Function) is calculated using the following formula:
  HOMA-Beta = [360 × Fasting insulin (μU/mL)] / [Fasting glucose (mg/dL) - 63]
  This approach evaluates the difference in beta-cell function changes across the groups over the study period, reflecting the intervention's impact on pancreatic function.
delta PSQI-BR scores (Pittsburgh Sleep Quality Index - Brazilian version) | 6, 12, 24 and 36 months
  To compare the mean delta PSQI-BR scores between groups:
  Delta = Mean PSQI-BR score at the final measurement - Mean PSQI-BR score at baseline
  The PSQI-BR (Pittsburgh Sleep Quality Index - Brazilian version) is a validated instrument used to assess sleep quality. It generates a total score based on seven components:
  Subjective sleep quality Sleep latency Sleep duration Habitual sleep efficiency Sleep disturbances Use of sleeping medications Daytime dysfunction Each component is scored from 0 to 3, and the total PSQI score ranges from 0 to 21, with higher scores indicating worse sleep quality.
  This approach evaluates the difference in sleep quality changes across the groups over the study period, reflecting the intervention's impact on sleep outcomes.
delta PSS-10 (Perceived Stress Scale - 10-item Brazilian version) | 6, 12, 24 and 36 months
  To compare the mean delta EPS-10 scores between groups:
  Delta = Mean EPS-10 score at the final measurement - Mean EPS-10 score at baseline
  The EPS-10 (Perceived Stress Scale - 10-item Brazilian version) is a validated instrument used to assess perceived stress over the last month. It consists of 10 questions scored on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often).
  The total score ranges from 0 to 40, with higher scores indicating greater perceived stress.
  This approach evaluates the difference in perceived stress levels across the groups over the study period, reflecting the intervention's impact on stress outcomes.
mean alcohol consumption (g/day) | 6, 12, 24 and 36 months
  To compare the mean alcohol consumption (g/day) between groups.
  Alcohol consumption will be assessed using a specific Alcohol Frequency Questionnaire, which records the type, frequency, and quantity of alcoholic beverages consumed. The total alcohol intake will be calculated in grams per day using the formula:
  Grams of alcohol/day = (Volume consumed [mL] × Alcohol content [%] × 0.8) / Days
  Where:
  Volume consumed is the reported quantity of alcoholic beverage. Alcohol content [%] is the average alcohol percentage for each beverage type. 0.8 is the density of pure ethanol.
  This approach evaluates changes in average daily alcohol consumption across the groups over the study period, reflecting the inter
  This approach evaluates the difference in perceived stress levels across the groups over the study period, reflecting the intervention's impact on stress outcomes.
proportion of smokers | 6, 12, 24 and 36 months
  To compare the proportion of smokers between groups at the end of the study:
  Smoking status will be assessed by self-report as either:
  Current smokers Former smokers Never smoked
  The proportion of smokers will be calculated as:
  Proportion of smokers (%) = (Number of smokers / Total participants in the group) × 100
  The comparison will focus on the proportion of current smokers in each group at the study's conclusion to evaluate the intervention's impact on smoking prevalence.
mean number of cigarettes smoked per day | 6, 12, 24 and 36 months
  To compare the mean number of cigarettes smoked per day between groups at the end of the study:
  Smoking behavior will be assessed by participants self-report the average number of cigarettes smoked per day.
  The mean number of cigarettes smoked per day for each group will be calculated as:
  Mean number of cigarettes/day = (Total number of cigarettes smoked by participants in the group) / (Number of participants who are current smokers)
  This comparison will evaluate the intervention's impact on the average smoking intensity among individuals who continue to smoke.
mean scores of the eight SF-36 quality of life domains | 6, 12, 24 and 36 months
  To compare the mean scores of the eight SF-36 quality of life domains between groups at the end of the study:
  Quality of life will be assessed using the SF-36 Health Survey, which evaluates eight domains:
  Physical functioning Role limitations due to physical health Role limitations due to emotional problems Energy/fatigue Emotional well-being Social functioning Pain General health
  Each domain generates a score ranging from 0 to 100, where higher scores indicate better quality of life.
  The mean scores for each domain will be calculated as:
  Mean domain score = (Sum of scores for all participants in the group) / (Number of participants in the group)
  This comparison will assess differences in quality of life between groups at the study's conclusion, reflecting the intervention's impact across various health dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Bersch-Ferreira, PhD, Principal Investigator — Hospital Beneficência Portuguesa de São Paulo
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Goiás - UFG, Goiânia, Goiás
  - Universidade Federal de Viçosa, Viçosa, Minas Gerais

IPD SHARING:
Plan to Share IPD: No